CLINICAL TRIAL: NCT01647945
Title: Single-Center Randomized Controlled Phase II Study of Safety and Efficacy of FK-506 (Tacrolimus) in Pulmonary Arterial Hypertension
Brief Title: FK506 (Tacrolimus) in Pulmonary Arterial Hypertension
Acronym: TransformPAH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Edda Spiekerkoetter (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor-Investigator, Edda Spiekerkoetter, Assistant Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAH-70522
Record Dates: First submitted 2012-07-18; First posted 2012-07-24 (Estimated); Results first posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH WHO group 1
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- FK506 level < 2 (Experimental)
  Interventions: Drug: FK506 level < 2 ng/ml
- FK506 level 2-3 (Experimental)
  Interventions: Drug: FK506 level 2-3 ng/ml
- FK506 level 3-5 (Experimental)
  Interventions: Drug: FK506 level 3-5 ng/ml

INTERVENTIONS:
Drug: Placebo — placebo pill
  Arms: Placebo
Drug: FK506 level < 2 ng/ml — FK506 goal trough blood level < 2 ng/ml
  Arms: FK506 level < 2
Drug: FK506 level 2-3 ng/ml — FK506 goal trough blood level 2-3 ng/ml
  Arms: FK506 level 2-3
Drug: FK506 level 3-5 ng/ml — FK506 goal trough blood level 3-5 ng/ml
  Arms: FK506 level 3-5

SUMMARY:
Mutations in bone morphogenetic protein receptor 2 (BMPR2) are present in >80% of familial and ~20% of sporadic pulmonary arterial hypertension (PAH) patients. Furthermore dysfunctional BMP signaling is a general feature of pulmonary hypertension even in non-familial PAH.

We therefore hypothesized that increasing BMP signaling might prevent and reverse the disease. We screened > 3500 FDA approved drugs for their propensity to increase BMP signaling and found FK506 (Tacrolimus) to be a strong activator of BMP signaling. Tacrolimus restored normal function of pulmonary artery endothelial cells, prevented and reversed experimental PAH in mice and rats.

Given that Tacrolimus is already FDA approved with a known side-effect profile, it is an ideal candidate drug to use in patients with pulmonary arterial hypertension.

The aims of our trial are:

1. Establish the Safety of FK506 in patients with PAH.
2. Evaluate the Efficacy of FK506 in PAH
3. Identify ideal candidates for future FK506 phase III clinical trial.

DETAILED DESCRIPTION:
Study Design:

Randomized, placebo-controlled, four arm clinical trial.

Sample Size: 10 subjects in each arm, Total enrollment = 40 patients.

1. 10 patients: FK-506 blood level: 3 - 5 ng/ml
2. 10 patients: FK-506 blood level: 2 - 3 ng/ml
3. 10 patients: FK-506 level: < 2.0 ng/ml
4. 10 patients: Placebo

Study Duration:

16 weeks

Primary Endpoints:

1) Safety of low-dose FK506 in PAH

Secondary Objectives/Endpoints:

1. Combined Clinical Events/Time to Clinical Worsening @ 16 weeks:

   * All cause mortality
   * Transplantation
   * Atrial septostomy
   * Need for escalation of therapies as deemed by site investigator
   * Worsening of NYHA/WHO classification by at least 1 point.
   * Hospitalization for right heart failure.
2. Change in 6MWD at 16 weeks
3. Change in NT-Pro-BNP at 16 weeks
4. Change in Uric Acid at 16 weeks
5. Change in DLCO at 16 weeks
6. Change in novel RV parameters by transthoracic echocardiography: Change in RV size, RA size, RV function, TAPSE, RVSP

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and < 70 years
2. Diagnosis of WHO Group I Pulmonary Arterial Hypertension (PAH) (Idiopathic (I)PAH, Heritable PAH (including Hereditary Hemorrhagic Telangiectasia), Associated (A)PAH (including collagen vascular disorders, drugs+toxins exposure, congenital heart disease, and portopulmonary disease).
3. Stable on active PAH treatment including any prostacycline or phosphodiesterase inhibitors and the endothelin antagonist Ambrisentan alone or in combination (stability defined as: <10% change in 6MWD, no change in NYHA class, no hospitalization or addition of PAH therapy for at least 3 months).
4. Previous Right Heart Catheterization that documented:

   1. Mean PAP ≥ 25 mmHg.
   2. Pulmonary capillary wedge pressure < 15 mmHg.
   3. Pulmonary Vascular Resistance ≥ 3.0 Wood units or 240 dynes/sec/cm5
5. WHO functional class I to IV as judged by the investigator.

Exclusion Criteria:

1. WHO Group II - V Pulmonary Hypertension.
2. Current or prior experimental PAH treatments within the last 6 months (including but not limited to tyrosine kinase inhibitors, rho-kinase inhibitors, or cGMP modulators).
3. Current active treatment with the dual endothelin receptor antagonist bosentan.
4. TLC < 60% predicted; if TLC b/w 60 and 70% predicted, high resolution computed tomography must be available to exclude significant interstitial lung disease.
5. FEV1 / FVC < 70% predicted and FEV1 < 60% predicted
6. Significant left-sided heart disease (based on screening Echocardiogram):

   1. Significant aortic or mitral valve disease
   2. Diastolic dysfunction ≥ Grade II
   3. LV systolic function < 45%
   4. Pericardial constriction
   5. Restrictive cardiomyopathy
   6. Significant coronary disease with demonstrable ischemia.
7. Chronic renal insufficiency defined as an estimated creatinine clearance < 30 ml/min (by MDRD equation).
8. Current atrial arrhythmias not under optimal control.
9. Uncontrolled systemic hypertension: SBP > 160 mm or DBP > 100mm
10. Severe hypotension: SBP < 80 mmHg.
11. Pregnant or breast-feeding.
12. Psychiatric, addictive, or other disorder that compromises patient's ability to provide informed consent, follow study protocol, and adhere to treatment instructions.
13. Active cyclosporine use.
14. Known allergy or hypersensitivity to FK-506.
15. Planned initiation of cardiac or pulmonary rehabilitation during period of study.
16. Human Immunodeficiency Virus infection.
17. Moderate to severe hepatic dysfunction with a Pugh score >10.
18. Hyperkalemia defined as Potassium > 5.1 mEq/L at screening .
19. Known active infection requiring antibiotic, antifungal, or antiviral therapies.
20. Co-morbid conditions that would impair a patient's exercise performance and ability to assess WHO functional class, including but not limited to chronic low-back pain or peripheral musculoskeletal problems.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edda Spiekerkoetter, MD, Principal Investigator — Stanford University; Roham Zamanian, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Derived] Spiekerkoetter E, Sung YK, Sudheendra D, Scott V, Del Rosario P, Bill M, Haddad F, Long-Boyle J, Hedlin H, Zamanian RT. Randomised placebo-controlled safety and tolerability trial of FK506 (tacrolimus) for pulmonary arterial hypertension. Eur Respir J. 2017 Sep 11;50(3):1602449. doi: 10.1183/13993003.02449-2016. Print 2017 Sep. PMID 28893866
- See also: Related Info — http://wallcenter.stanford.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | FK506 Level < 2 | FK506 Level 2-3 | FK506 Level 3-5
Started | 6 | 6 | 5 | 6
Completed | 6 | 6 | 3 | 5
Not Completed | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | FK506 Level < 2 | FK506 Level 2-3 | FK506 Level 3-5 | Total
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 5 | 6 | 23
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46 [38 to 53] | 35 [24 to 45] | 39 [25 to 51] | 45 [42 to 48] | 41 [34 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 3 | 4 | 16
  Male | 1 | 2 | 2 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 5 | 6 | 23

OUTCOME MEASURES:

1. Primary Outcome: Safety of Low-dose FK-506 in PAH
Description: Total number of adverse events measured between baseline and end of study at 18 weeks as reported by study subjects such as nausea/diarrhea, URI, sinus congestion, infection, fluid retention/edema, cough, headache, bronchitis, fatigue, drug reaction/hives, flushing, anxiety, tremor, fever, shingles, SOB, insomnia, pain
Time Frame: 18 weeks
Population: all study subjects who started the study
Measure: Number; unit: number of AEs
Arm/Group | Placebo | FK506 Level < 2 | FK506 Level 2-3 | FK506 Level 3-5
Number analyzed (Participants) | 6 | 6 | 5 | 6
number of AEs | 8 | 18 | 9 | 22

2. Secondary Outcome: Number of Combined Clinical Events
Description: Combined Clinical Events @ 16 weeks:
  Number of patients who died Number of patients who got transplanted Number of patients who needed escalation of therapies Number of patients who had worsening of NYHA/WHO classification by at least 1 point Number of patients who require hospitalization for right heart failure
  Low numbers would suggest either efficacy of the study drug or slowly progression of disease that is studied during the 16 week study period or short observation period or small study population
Time Frame: Baseline to 16 weeks
Population: Subjects were included who finished the 16 week study period. A total of 3 participants did not complete the study
Measure: Number; unit: Combined Number of Clinical Events
Arm/Group | Placebo | FK506 Level < 2 | FK506 Level 2-3 | FK506 Level 3-5
Number analyzed (Participants) | 6 | 6 | 3 | 5
Combined Number of Clinical Events | 0 | 0 | 0 | 0

3. Secondary Outcome: Efficacy of Low-dose FK-506 in Pulmonary Arterial Hypertension (PAH) Measured by Change in 6-min Walk Distance (6MWD)
Description: Change in 6MWD in meter between baseline and 16 weeks
  A large number would indicate an increase in exercise capacity
Time Frame: baseline to 16 weeks
Population: Only subjects were included who finished the 16-week study 3 patients did not finish
Measure: Median (Inter-Quartile Range); unit: meter
Arm/Group | Placebo | FK506 Level < 2 | FK506 Level 2-3 | FK506 Level 3-5
Number analyzed (Participants) | 6 | 6 | 3 | 5
meter | 14.5 [3.5 to 38.25] | 0 [-20.25 to 3] | 41 [-9.5 to 59] | 0 [-20 to 9]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from every study subject who started the study regardless whether the subject finished the study. Events were collected during the time frame between baseline and 18 weeks.
Description: Of note the study drug was stopped at 16 weeks, an additional observation period of 2 weeks was used to capture possible adverse events of study drug.
Arm/Group | Placebo | FK506 Level < 2 | FK506 Level 2-3 | FK506 Level 3-5
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 6/6 | 4/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | FK506 Level < 2 (N=6) | FK506 Level 2-3 (N=5) | FK506 Level 3-5 (N=6)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — One patient developed hemoptysis during the observation weeks 16 -18, after the study drug had already been stopped (at week 16). The hemoptysis occured in the setting of a strep throat infection that was treated with antibiotics.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | FK506 Level < 2 (N=6) | FK506 Level 2-3 (N=5) | FK506 Level 3-5 (N=6)
Nausea/ Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 5 (6)
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4) | 0 (0) | 1 (1)
Sinus congestion (General disorders) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fluid retention (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) — not requiring increase in diuretics

LIMITATIONS AND CAVEATS:
Due to slow patient recruitment in single academic center we recruited fewer patients than originally expected.

Follow-up multicenter phase IIb efficacy trial is planned

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes